CLINICAL TRIAL: NCT04797949
Title: Adherence to Universal Aspirin Compared to Screening Indicated Aspirin for Prevention of Preeclampsia
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Sebastian Ramos, Principal Investigator, Women and Infants Hospital of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1581227
Record Dates: First submitted 2021-02-08; First posted 2021-03-15 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Medication Adherence; Preeclampsia
Keywords: aspirin; preeclampsia; adherence; pregnancy
MeSH Terms: conditions — Medication Adherence; Pre-Eclampsia | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Patients are randomized to receiving aspirin knowing their risk status vs those who are randomized to universal receipt.
Who Masked: Outcomes Assessor
Masking Description: The study personnel who will perform pill counts will be masked to the study arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Randomized to USPSTF Criteria (Active Comparator): Women randomized to knowing their risk of preeclampsia and therefore, candidates for low dose aspirin.
  Interventions: Drug: Low-dose aspirin
- Randomized to Universal aspirin receipt (Active Comparator): Women randomized to receiving low dose aspirin without knowing their risk status.
  Interventions: Drug: Low-dose aspirin

INTERVENTIONS:
Drug: Low-dose aspirin — Women will be prescribed 81 mg of aspirin to take daily during pregnancy.

SUMMARY:
There are data showing that a majority of pregnant women may not be accurately identified as high risk through screening and therefore, not receiving prophylactic low dose aspirin as recommended. This leads to missing many patients who would benefit from aspirin administration. Aspirin is an effective, affordable and safe intervention and its universal use in pregnancy has been proposed as the answer to help mitigate risk of significant morbidity from preeclampsia. However, adherence to aspirin in women at low risk compared to those deemed at high risk of preeclampsia has never been studied. One of the arguments against universal aspirin administration is the concern that universal receipt would change the compliance in those at high risk although there are no data to support this concern. To address the lack of data on differences in adherence, our goal in this proposal is to assess whether there is a difference in adherence to low dose aspirin (81 mg) in women at high risk of preeclampsia as indicated by USPSTF risk algorithm when compared to those women randomized to universal use.

DETAILED DESCRIPTION:
Research objective- To compare adherence to low dose, 81mg of aspirin in women considered high risk by USPSTF criteria vs universal receipt.

Hypothesis: Women considered high risk by USPSTF criteria will have better adherence to low dose aspirin than women randomized to universal receipt.

Study Design: Randomized trial

Population: English or Spanish speaking women between 10-20 weeks of gestation receiving their care at Women & Infants Hospital, with a plan to deliver at Women & Infants Hospital

Once enrolled, patients will then be randomized to USPSTF criteria to determine if they qualify for aspirin or to universal aspirin receipt. Once randomized, patients will undergo video pill counts at multiple intervals in their prenatal care (monthly).

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 10 to 20 weeks gestation by best available dating
* 18 years of age or older
* Fluency in English or Spanish

Exclusion Criteria:

• Contraindication to aspirin use

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only pregnant individuals will be included regardless of gender identity.
Enrollment: 0 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to aspirin use | up to 42 weeks.
  A Research Coordinator will contact each patient within 7 days of recruitment to assure the patient has picked up and has their prescription with subsequent contacts occurring at 30-day intervals until delivery.

SECONDARY OUTCOMES:
Rates of postpartum hemorrhage | These will be assessed within 24 hours after delivery.
  We will collect information at time of delivery of rates of postpartum hemorrhage defined as estimated blood loss of 1000 cc or greater.
Rates of preeclampsia | Rates of hypertensive disease of pregnancy will be measured from 20 weeks of gestation until 6 weeks postpartum
  We will measure rates of hypertensive disease of pregnancy
Fetal growth restriction | This will be measured from 24 weeks until 39 weeks.
  We will measure rates of fetal growth restriction defined as estimated fetal weight or abdominal circumference <10%ile.
Placental abruption | This will be measured from 20 weeks until 42 weeks.
  Rates of placental abruption will be collected

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Z Ramos, MD, Principal Investigator — Women and Infants Hospital
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Ayala NK, Rouse DJ. A Nudge Toward Universal Aspirin for Preeclampsia Prevention. Obstet Gynecol. 2019 Apr;133(4):725-728. doi: 10.1097/AOG.0000000000003167. PMID 30870274
- [Result] Mone F, Mulcahy C, McParland P, Breathnach F, Downey P, McCormack D, Culliton M, Stanton A, Cody F, Morrison JJ, Daly S, Higgins J, Cotter A, Hunter A, Tully EC, Dicker P, Alfirevic Z, Malone FD, McAuliffe FM. Trial of feasibility and acceptability of routine low-dose aspirin versus Early Screening Test indicated aspirin for pre-eclampsia prevention (TEST study): a multicentre randomised controlled trial. BMJ Open. 2018 Jul 28;8(7):e022056. doi: 10.1136/bmjopen-2018-022056. PMID 30056389
- [Result] Shanmugalingam R, Wang X, Motum P, Fulcher I, Lee G, Kumar R, Hennessy A, Makris A. Clinical Influence of Nonadherence With Prophylactic Aspirin in Preventing Preeclampsia in High-Risk Pregnancies: A Multicenter, Prospective, Observational Cohort Study. Hypertension. 2020 Apr;75(4):1125-1132. doi: 10.1161/HYPERTENSIONAHA.119.14107. Epub 2020 Mar 2. PMID 32114852
- [Result] Werner EF, Hauspurg AK, Rouse DJ. A Cost-Benefit Analysis of Low-Dose Aspirin Prophylaxis for the Prevention of Preeclampsia in the United States. Obstet Gynecol. 2015 Dec;126(6):1242-1250. doi: 10.1097/AOG.0000000000001115. PMID 26551178
- [Result] Henderson JT, Whitlock EP, O'Connor E, Senger CA, Thompson JH, Rowland MG. Low-dose aspirin for prevention of morbidity and mortality from preeclampsia: a systematic evidence review for the U.S. Preventive Services Task Force. Ann Intern Med. 2014 May 20;160(10):695-703. doi: 10.7326/M13-2844. PMID 24711050